CLINICAL TRIAL: NCT03516539
Title: Comparison of the Mcgrath Videolaryngoscope With the Macintosh Laryngoscope for Orotracheal Intubation in Patients With Manual In-line Stabilization
Brief Title: Mcgrath Videolaryngoscope Versus Macintosh Laryngoscope in Patients With Manual In-line Stabilization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-I043
Record Dates: First submitted 2018-04-24; First posted 2018-05-04 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-04

CONDITIONS: Anesthesia, General
Keywords: Videolaryngoscopy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ML (Experimental): Mcgrath videolaryngoscopy
  Interventions: Device: Group ML
- Group DL (Active Comparator): direct Macintosh laryngoscope
  Interventions: Device: Group DL

INTERVENTIONS:
Device: Group ML — Mcgrath videolaryngoscope
  Arms: Group ML
Device: Group DL — Macintosh laryngoscope
  Arms: Group DL

SUMMARY:
Video laryngoscopy provides easily a good laryngeal view compared to direct laryngoscopy. It is particularly, useful in patients with anticipated difficult intubation, and also widely used for educational purposes. Among video laryngoscopy, Mcgrath is a recently-developed, portable video laryngoscopy with a liquid crystal display (LCD) monitor and disposable curved blade.

Mcgrath is known to provide excellent laryngeal visibility even in case of anticipated-difficult and anticipated-unsuccessful intubation as well as normal airway management. However, compared with direct laryngoscopy, the success rate of intubation and the time required for anticipated difficult intubation have been reported conflicting results in previous studies. The aim of this study was to compare the intubation success rate, the intubation time and the ease of use with Mcgrath video laryngoscopy and direct laryngoscopy during intubation.

DETAILED DESCRIPTION:
1. In the operating room, all patients are monitored with an electrocardiograph, noninvasive blood pressure, pulse oximeter, capnograph and Bispectral index (BIS) monitor. After pre-oxygenation with 100% oxygen for 1 minute, intravenous anesthesia (TIVA) with propofol and remifentanyl is administrated and followed by rocuronium (0.6mg/kg). When patients are lost their consciousness, manual mask ventilation is proceeded with 100% oxygen for 2 minutes.
2. Transoral endotracheal intubation is performed using Mcgrath videolaryngoscope (Group ML) and direct laryngoscope (Group DL) using manual in-line stabilization. At this time, the time required for intubation is measure by other medical personnel not engaged in this research.
3. The anesthesiologist assesses Cormack Lehane laryngeal visual field,external laryngeal manipulation, intubation difficulty scales (IDS) and the difficulty of intubation.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for general anesthesia requiring tracheal intubation. Patients are aged 19 to 70 years and are American Society of Anesthesiologists physical status I, II.

Exclusion Criteria:

* Patients requiring rapid sequence intubation Patients with poor teeth or high risk of aspiration pneumonia Cervical spine pathology, pharyngeal pathology

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-12-11 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-07-07 (Estimated)

PRIMARY OUTCOMES:
Intubation success rate | 1 hour
  success or failure of intubation

SECONDARY OUTCOMES:
Time required for intubation | 1 hour
  time until end tidal carbon dioxide (CO2) measurement after laryngeal blade passing through patient's teeth
Intubation difficulty score | 1 hour
  difficulty at the time of intubation. (easy /moderate/ difficult)
Complications | 1 day
  oral bleeding, teeth or lip bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Yi Hwa Choi, Dr, Study Director — Halllym university Sacred Hospital
Locations (1):
- Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rai MR, Dering A, Verghese C. The Glidescope system: a clinical assessment of performance. Anaesthesia. 2005 Jan;60(1):60-4. doi: 10.1111/j.1365-2044.2004.04013.x. PMID 15601274
- [Background] Asai T, Murao K, Shingu K. Training method of applying pressure on the neck for laryngoscopy: use of a videolaryngoscope. Anaesthesia. 2003 Jun;58(6):602-3. doi: 10.1046/j.1365-2044.2003.03207_7.x. No abstract available. PMID 12846635
- [Result] Shippey B, Ray D, McKeown D. Case series: the McGrath videolaryngoscope--an initial clinical evaluation. Can J Anaesth. 2007 Apr;54(4):307-13. doi: 10.1007/BF03022777. PMID 17400984
- [Result] Shippey B, Ray D, McKeown D. Use of the McGrath videolaryngoscope in the management of difficult and failed tracheal intubation. Br J Anaesth. 2008 Jan;100(1):116-9. doi: 10.1093/bja/aem303. Epub 2007 Oct 23. PMID 17959584